CLINICAL TRIAL: NCT00231803
Title: Canadian Collaborative Group for the Prevention of Illness in Chronic Renal Disease: The Canadian Prevention of Renal and Cardiovascular Endpoints Trial
Brief Title: The Canadian Prevention of Renal and Cardiovascular Endpoints Trial
Acronym: CanPrevent
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brendan Barrett (Other)
Collaborators: Nova Scotia Health Authority (Other); Hopital Charles Lemoyne (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); University of British Columbia (Other)
Responsible Party: Sponsor-Investigator, Brendan Barrett, Professor of Medicine, Memorial University of Newfoundland
Organization: Memorial University of Newfoundland (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HIC#04.154
Record Dates: First submitted 2005-09-30; First posted 2005-10-04 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Chronic Kidney Disease
Keywords: Cardiovascular; Prevention; RCT
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multifactorial intervention (Experimental): Nurse led clinic involving a nephrologist administering protocol driven interventions aimed at preservation of kidney function, and cardiovascular risk reduction. Blood pressure targets were specified. No specific drugs were specified. Drug classes such as primarily statins for achieving LDL targets, use of an ACE inhibitor or ARB if possible, treatment of acidosis, anemia, hyperphosphatemia, advice on smoking cessation
  Interventions: Other: Combined CKD and CVD Prevention; Other: Cardiovascular Disease prevention; Other: Treatment of Chronic Kidney Disease complications
- Usual care (Active Comparator): Usual care includes any intervention thought appropriate by the treating family doctor and or specialists involved in the case
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Combined CKD and CVD Prevention — Perindopril, Lisinopril, Captopril, Candesartan, Losartan, Amlodipine, Verapamil, Chlorthalidone
  Arms: Multifactorial intervention
Other: Cardiovascular Disease prevention — Atorvastatin, Rosuvastatin, Simvastatin, Aspirin, Clopidogrel
  Arms: Multifactorial intervention
Other: Treatment of Chronic Kidney Disease complications — Calcitriol, Calcium carbonate, Erythropoietin, Sodium bicarbonate
  Arms: Multifactorial intervention
Other: Usual care — No prescribed intervention, just those that the patient's own family physician thought indicated
  Arms: Usual care

SUMMARY:
Advanced kidney disease with it's associated heart and blood vessel problems are becoming more frequent. These problems markedly affect length and quality of life and cost a lot to treat. Treatments are known that can prevent development of advanced kidney and heart disease. These treatments are not being optimally applied in the current health system. This study aims to identify people with relatively early stage chronic kidney disease. With the participation of these people, the study will test whether a nurse coordinated clinic involving a medical kidney specialist, applying the known treatments, can reduce or delay the onset of advanced kidney disease and heart and blood vessel problems such as heart attack, stroke and death, to a greater extent than usual care. The study will also address issues of costs associated with care and illness. The nature of the care provided by the health care professionals will be studied to see how best to achieve good health outcomes.

DETAILED DESCRIPTION:
The pilot study is designed in two phases. The first phase is intended to provide data on some key points that need to be addressed prior to future funding applications to the CIHR and the NHLBI. These applications are currently tentatively planned for the fall of 2005. The second phase of the pilot study is intended to more completely establish the feasibility of successfully completing the full trial by examining the issue of contamination and the ability of the intervention to generate a difference between the groups with regard to use of efficacious therapies and control of modifiable risk factors, or intermediate variables on the causal pathway to the clinical end-points in the full-scale trial. The second phase will also address the need to describe the operation of the experimental intervention more thoroughly. Finally, the second phase of the pilot study will compare the randomized study groups with regard to short-term quality-of-life outcomes.

Phase1

1. How long does it take to recruit 100 patients per study site?
2. What recruitment strategies are most efficient?
3. How do the baseline characteristics of those recruited compare to referred populations, and to the general population with CKD?
4. How do the nephrologist and nurse work together to provide care to those in the intervention group?
5. What is the nature of the care provided by the nurses and physicians to those in the intervention group?
6. Is the study nurse able to manage the patient load?
7. How much time and resources are needed to a) provide care, b) to carry out study measurements?
8. Can health care resources used be measured for economic analysis?

Phase II

1. What is the rate of loss to follow-up?
2. What is the overall estimate of the primary outcome event rate?
3. By one year of follow-up, what is the difference between the study groups in terms of:

   1. Protocol interventions used (estimates contamination)
   2. Proportion i) smoking; and proportion achieving ii) BP, iii) lipid, iv) diabetes, v) anemia, vi) acidosis, vii) mineral metabolism targets
   3. Quality of Life
   4. Satisfaction with care Randomized, parallel, two group, multicentre, clinical trial of people with CKD, with or without diabetes mellitus or proteinuria. The intention is to roll the pilot study into the full-scale trial if the pilot itself is deemed successful. A laboratory-based case finding method will be used preferentially to identify potential participants. This will be supplemented by practice-based case-finding approaches where necessary to ensure recruitment of a representative population. Randomization will be by a central computer-based telephone process. Stratification will be by center and presence of diabetes and proteinuria. The intervention consists of a protocol guided, multiple risk factor and chronic disease care model-like approach delivered by a trained nurse supported by a nephrologist and will be based in a nephrology clinic like setting.

ELIGIBILITY:
Inclusion Criteria:

* Stratum 1 (expected about 50% of trial subjects): Diabetes mellitus (by clinical history with documented prior plasma glucose levels in the diabetic range, or on hypoglycemic medications) and CKD as documented by calculated (Cockroft-Gault equation) creatinine clearance between 25 and 60 mls/min/1.73m2 derived from the screening serum creatinine value and the next most recent known value from more than 2 weeks prior; OR

Stratum 2 (expected about 20% of trial subjects): Non-diabetic with CKD as defined for Stratum 1 and proteinuria of > 1g/L by dipstick in random urine at screening; OR

Stratum 3 (expected about 30% of trial subjects): Non-diabetic with CKD as defined for stratum 1, but without proteinuria as for stratum 2 at screening

Exclusion Criteria:

* Unwilling to provide informed consent
* Likely to die of any known existing disease within 6 months
* Recently unstable/advanced cardiovascular disease (MI or acute coronary syndrome, hospitalized heart failure, TIA or stroke, leg amputation or gangrene in past 6 months)
* Currently receiving active treatment for a malignant, neoplastic disease other than localized non-melanoma skin cancer
* Progressive kidney disease currently treated by immunotherapy
* Currently receiving dialysis or likely to do so within 6 months
* Current organ transplant recipient (or planned within 6 months)
* Currently receiving ongoing care for CKD, or cardiovascular disease, in a multiple intervention, disease management program.
* Currently enrolled in another interventional trial
* Residing in a location not amenable to follow up for the trial

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Actual)
Dates: Start 2005-04; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Time to major cardiovascular event(myocardial infarction, stroke, coronary or peripheral revascularization, hospitalization for heart failure or unstable angina, or death due to cardiovascular cause) | 24 months
  Blind expert panel determined major cardiovascular events or death
Time to first major clinical event (ESRD, non-fatal cardiovascular events as in secondary (a) or all cause death) | 24 months
  Blind expert panel determined major cardiovascular event, death or end stage renal disease

CONTACTS AND LOCATIONS:
Overall Officials: Patrick S Parfrey, MD, Principal Investigator — Memorial University of Newfoundland; Brendan J Barrett, MD, Principal Investigator — Memorial University of Newfoundland
Locations (5):
- Canada (5):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Memorial University of Newfoundland, St. John's, Newfoundland and Labrador
  - Capitol District Health Authority, Halifax, Nova Scotia
  - London Health Sciences Centre, London, Ontario
  - Charles LeMoyne Hospital, Greenfield Park, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Publication of study design and results in open access
Supporting Information: Study Protocol, CSR
Time Frame: by 2011
Access Criteria: Indefinite
URL: https://pubmed.ncbi.nlm.nih.gov/21617090/

REFERENCES:
- [Derived] Hopkins RB, Garg AX, Levin A, Molzahn A, Rigatto C, Singer J, Soltys G, Soroka S, Parfrey PS, Barrett BJ, Goeree R. Cost-effectiveness analysis of a randomized trial comparing care models for chronic kidney disease. Clin J Am Soc Nephrol. 2011 Jun;6(6):1248-57. doi: 10.2215/CJN.07180810. Epub 2011 May 26. PMID 21617091
- [Derived] Barrett BJ, Garg AX, Goeree R, Levin A, Molzahn A, Rigatto C, Singer J, Soltys G, Soroka S, Ayers D, Parfrey PS. A nurse-coordinated model of care versus usual care for stage 3/4 chronic kidney disease in the community: a randomized controlled trial. Clin J Am Soc Nephrol. 2011 Jun;6(6):1241-7. doi: 10.2215/CJN.07160810. Epub 2011 May 26. PMID 21617090